CLINICAL TRIAL: NCT00135876
Title: A Trial of Dalteparin Low Molecular Weight Heparin for Primary Prophylaxis of Venous Thromboembolism in Brain Tumour Patients (PRODIGE)
Brief Title: Dalteparin Low Molecular Weight Heparin for Primary Prophylaxis of Venous Thromboembolism in Brain Tumour Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 524E-CVD-0056-013
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Venous Thromboembolism; Brain Tumors
Keywords: deep vein thrombosis; pulmonary embolism; glioma; fragmin; anticoagulant; prophylaxis; dalteparin
MeSH Terms: conditions — Venous Thromboembolism; Brain Neoplasms; Venous Thrombosis; Pulmonary Embolism; Glioma | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dalteparin

SUMMARY:
In patients with malignant glioma, to determine the efficacy of prophylaxis with LMWH (dalteparin) compared to placebo, both commenced beyond the immediate postoperative period, for the prevention of VTE.

DETAILED DESCRIPTION:
Patients are randomized 1:1 to receive dalteparin 5,000 anti-Xa units s.c. daily versus placebo s.c. daily. The primary outcome is VTE-free survival at 6 months. Progression free survival; overall survival, toxicity, and neurocognitive performance are secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Both of the following criteria must be satisfied:

  1. Patients with newly-diagnosed pathologically-confirmed WHO Grade 3 or Grade 4 glioma (anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic oligodendroglioma, and anaplastic mixed glioma). Tumour histology is based on local pathology review only;
  2. Patients 18 years of age or older at time of randomization

Exclusion Criteria:

* If one or more of the following criteria are satisfied, the patient is not eligible for the study:

  1. The presence of acute or chronic DVT demonstrated by duplex ultrasonography (DUS) or venography. (Note: a screening DUS is not required for study entry);
  2. Inability to commence study drug within four weeks of original surgery or biopsy;
  3. Serious hemorrhage requiring hospitalization, transfusion, or surgical intervention within four weeks of potential study entry;
  4. Presence of a coagulopathy (e.g. INR >1.5 or platelet count < 100x109/L);
  5. Symptomatic intracranial or intratumoural bleeding. (Note: post-operative imaging of the brain is not required for study entry. Asymptomatic "routine" post-operative blood products in a post-surgical cavity are not an exclusion;
  6. Known acute (symptomatic or actively bleeding) gastroduodenal ulcer;
  7. Familial bleeding diathesis;
  8. Requiring long term anticoagulants for other reasons (e.g., mechanical heart valves, atrial fibrillation);
  9. Uncontrolled hypertension despite antihypertensive therapy;
  10. Significant renal failure (dependent on dialysis or creatinine of greater than three times upper limit of normal control);
  11. Prior history of documented DVT or PE;
  12. Allergy to anticoagulants (UFH, LMWH) including immune-mediated heparin-induced thrombocytopenia;
  13. Pregnant or of childbearing potential and not using adequate contraception;
  14. Geographically inaccessible for follow-up;
  15. Having an expected life span of less than 6 months;
  16. Body weight < 40 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512
Dates: Start 2002-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
objectively-proven symptomatic VTE (DVT or PE)

SECONDARY OUTCOMES:
bleeding (major and all bleeding)
quality of life
cognition assessments
death

CONTACTS AND LOCATIONS:
Overall Officials: James Perry, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); William Geerts, MD, Principal Investigator — Toronto Sunnybrook Regional Cancer Centre; Jim Julian, MMath, Principal Investigator — McMaster University, Dept of Clinical Epidemiology & Biostatistics
Locations (14):
- United States (3):
  - Kellogg Cancer Center - Evanston Northwestern Healthcare, Evanston, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (3):
  - The St. George Hospital, Kogarah, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Toronto-Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Italy (2):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Università di Perugia, Perugia